CLINICAL TRIAL: NCT05925270
Title: Substituting SMSs for Provider-delivered Care to Improve Alcohol Use Outcomes in People With and Without HIV in Lesotho
Brief Title: Substituting SMSs for Provider-delivered Care to Improve Alcohol Use Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: SolidarMed (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID02-2023; U1111-1292-9288 (Other: World Health Organization)
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder, Mild; Alcohol Use Disorder, Moderate
Keywords: SMSs; alcohol use; Mental Health Gap Action Programme (mhGAP); Lesotho
MeSH Terms: conditions — Alcoholism; Lymphoma, Follicular; Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mhGAP-Remote (Experimental): mhGAP-Remote was developed specifically by our team. It involves the same intervention components described in mhGAP-Standard. However, in mhGAP-Remote the intervention is delivered mostly through standardized SMSs. There is one in-person session with the interventionist, where the participant learns the core skills of mhGAP. This is followed by standardized SMSs to reinforce intervention content learned in the first session. Study interventionists will be able to provide brief telephonic support to participants if participants struggle to implement the skills learned.
  Interventions: Behavioral: mhGAP-Remote
- mhGAP-Standard (Active Comparator): mhGAP-Standard refers to the existing evidence-based intervention guide that was developed by the WHO to help non-specialist providers in LMIC settings provide treatment for alcohol use, among other mental health and neurological conditions. For the current study, the intervention will focus on mhGAP's psychosocial interventions, which involve psychoeducation, brief motivational interviewing, and providing strategies to reduce and/or stop use. The intervention uses a harm reduction approach, meaning that participants do not need to stop using alcohol altogether. Interventionists will deliver 4 sessions, approximately 45-60 mins each, to participants in person. Sessions are designed to be delivered approximately weekly. Providers have the option to deliver up to 2 additional "booster sessions" to participants who may benefit from additional care.
  Interventions: Behavioral: mhGAP-Standard

INTERVENTIONS:
Behavioral: mhGAP-Remote — One in-person session followed by standardized SMSs to reinforce the concepts learned in the first session. The intervention follows principles of the World Health Organization's Mental Health Gap Action Programme (mhGAP). Study interventionists can provide telephonic support to participants to implement the skills.
  Arms: mhGAP-Remote
Behavioral: mhGAP-Standard — Four in-person sessions with up to two booster sessions following the principles of World Health Organization's Mental Health Gap Action Programme (mhGAP).
  Arms: mhGAP-Standard

SUMMARY:
The goal of this clinical trial is to test whether a technology-substituted intervention (mhGAP-Remote) derived from the World Health Organization's (WHO) Mental Health Gap Action Programme-Intervention Guide (mhGAP-IG) is effective to reduce alcohol use among adults with and without HIV in Lesotho. Participants who receive the mhGAP-Remote intervention will complete one in-person intervention session pertaining to the mhGAP-IG module for alcohol use, followed by short message services (SMSs) related to the intervention material covered during the in person session. This will be compared to mhGAP-Standard, which involves 4 in-person sessions based on mhGAP-IG for alcohol use plus the option of 2 additional booster sessions. Participants in both treatment groups will complete assessments at baseline, 8-weeks follow-up, 20-weeks follow-up, and 32-weeks follow-up, consisting of self-reported questionnaires and laboratory tests.

DETAILED DESCRIPTION:
Mental health and alcohol and other drug use problems account for over 20% of the years lived with disability globally, including in low- and middle-income countries (LMICs). Unfortunately, there is a severe shortage of treatment providers available in LMICs for these problems, and access to care is limited due to cost, transportation, infrastructure, lack of awareness, and stigma. The use of technology as a substitute for some provider-delivered time is an appealing and promising strategy to increase access to alcohol use treatment. Specifically, using SMSs to deliver intervention content is a feasible approach in low-resource settings and has been successfully implemented for other behavioral health problems. The primary objective of this study is to test the effectiveness of a technology substituted mhGAP intervention, mhGAP-Remote, to reduce alcohol use when compared to standard in-person treatment, mhGAP-Standard. Study results can inform barriers to accessing treatment and care for alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Meets criteria for "hazardous drinking" according to the AUDIT (total score of ≥ 6 for women, ≥ 8 for men)
* Has cellphone access at least half the days of the week, regular access to electricity to charge the phone, and is comfortable receiving study-specific SMSs related to alcohol use treatment on the phone
* Willing to participate in a study focused on problem drinking
* Willing and able to regularly come to the health facility/clinic for intervention sessions during the active intervention period
* Able to read in Sesotho or English or has a treatment supporter (e.g., family member) able to read study-related materials
* Willing to have intervention sessions audio-recorded
* Attends one of the study clinics and intends to remain at the same clinic for the duration of the trial

Exclusion Criteria:

* High-risk alcohol use that warrants medical management
* Known brain tumor or brain damage, history of epilepsy, or history of delirium
* Untreated major mental illness that interferes with study participation, such as psychosis, or mania
* Reported pregnancy at time of enrolment
* Currently receiving psychological treatment for alcohol use
* Participation in another trial that is judged by the site investigator as non-compatible with this study
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Self-reported alcohol use | Change from baseline to approximately 8-weeks follow-up [range 6--16 weeks]
  Self-report using the Alcohol Use Disorder Identification Test (AUDIT). Higher scores indicate more alcohol use and associated problems.

SECONDARY OUTCOMES:
Self-reported alcohol use | Change from baseline to approximately 20-weeks [range >16--28 weeks] and 32-weeks follow-up [range >28--40 weeks]
  Self-report using the Alcohol Use Disorder Identification Test (AUDIT). Higher scores indicate more alcohol use and associated problems.
Biomarker phosphatidylethanol (PEth) | Change from baseline to approximately 8-weeks [range 6--16 weeks], 20-weeks [range >16--28 weeks], and 32-weeks follow-up [range >28--40 weeks]
  PEth concentration in dried blood spots

OTHER OUTCOMES:
HIV viral load | Change from baseline to approximately 8-weeks [range 6--16 weeks], 20-weeks [range >16--28 weeks], and 32-weeks follow-up [range >28--40 weeks]
  For patients with HIV, number of copies of HIV per millimeter in dried blood spots
Liver function | Change from baseline to approximately 8-weeks [range 6--16 weeks], 20-weeks [range >16--28 weeks], and 32-weeks follow-up [range >28--40 weeks]
  Aspartate Aminotransferase and Alanine Aminotransferase in whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M. Belus, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (3):
- Lesotho (3):
  - Butha Buthe District Hospital, Butha-Buthe, Butha-Buthe
  - Seboche Hospital, Butha-Buthe, Butha-Buthe
  - St. Paul's Health Centre, Butha-Buthe, Butha-Buthe

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized data and statistical code will be deposited alongside the published peer-reviewed papers, in alignment with data sharing and verification procedures. Other investigators wishing to access the data for additional analyses can contact the study PI so that the appropriate documents (e.g., data sharing, ethics approvals) can be arranged.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: A de-identified dataset will be deposited in an open-access data repository at the end of the project and once the objectives specified in the protocol have been addressed.
Access Criteria: The data can be accessed by the public, through creation of an account with Open Science Foundation, an open-access data repository.
URL: https://osf.io/ftqyd/

REFERENCES:
- [Background] Campbell AN, Nunes EV, Matthews AG, Stitzer M, Miele GM, Polsky D, Turrigiano E, Walters S, McClure EA, Kyle TL, Wahle A, Van Veldhuisen P, Goldman B, Babcock D, Stabile PQ, Winhusen T, Ghitza UE. Internet-delivered treatment for substance abuse: a multisite randomized controlled trial. Am J Psychiatry. 2014 Jun;171(6):683-90. doi: 10.1176/appi.ajp.2014.13081055. PMID 24700332
- [Background] Hahn JA, Dobkin LM, Mayanja B, Emenyonu NI, Kigozi IM, Shiboski S, Bangsberg DR, Gnann H, Weinmann W, Wurst FM. Phosphatidylethanol (PEth) as a biomarker of alcohol consumption in HIV-positive patients in sub-Saharan Africa. Alcohol Clin Exp Res. 2012 May;36(5):854-62. doi: 10.1111/j.1530-0277.2011.01669.x. Epub 2011 Dec 7. PMID 22150449
- [Background] mhGAP Intervention Guide for Mental, Neurological and Substance Use Disorders in Non-Specialized Health Settings: Mental Health Gap Action Programme (mhGAP). Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138690/ PMID 23741783
- [Background] Atkins DL, Cumbe VFJ, Muanido A, Manaca N, Fumo H, Chiruca P, Hicks L, Wagenaar BH. Validity and item response theory properties of the Alcohol Use Disorders Identification Test for primary care alcohol use screening in Mozambique (AUDIT-MZ). J Subst Abuse Treat. 2021 Aug;127:108441. doi: 10.1016/j.jsat.2021.108441. Epub 2021 Apr 28. PMID 34134876
- [Derived] Belus JM, Johnson NE, Yoon GH, Tschumi N, Lerotholi M, Falgas-Bague I, Lee TT, Letsoela P, Magidson JF, Amstutz A, Labhardt ND. SMSs as an alternative to provider-delivered care for unhealthy alcohol use: study protocol for Leseli, an open-label randomised controlled trial of mhGAP-Remote vs mhGAP-Standard in Lesotho. Trials. 2024 Sep 2;25(1):575. doi: 10.1186/s13063-024-08411-3. PMID 39223600